CLINICAL TRIAL: NCT04885959
Title: The Effects of Traditional Asian Diet on Gut Microbiome and Metabolome in Healthy Volunteers and Pregnancy on Subsequent Infant's Allergy Development
Brief Title: Traditional Asian Diet and Gut Microbiome and Metabolome in Healthy Volunteers and Pregnancy on Infant's Allergy Development
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Nur-Fazimah Sahran, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: USM/JEPeM/20120611
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy; Food Hypersensitivity; Healthy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual diet (No Intervention): In the pilot study among healthy volunteers, participant need to maintain their habitual diet for 4 weeks. Meanwhile, in the large-scale study among pregnant women, participants are subjected to receive general dietary advice for healthy pregnancy from attended nurses or physician during their antenatal visits.
- Traditional Asian Diet (Experimental): Participants will receive dietary intervention on a traditional Asian diet which diet consists of high fiber, moderate protein, and low fat and with the inclusion of local probiotics and prebiotics food sources which are known to enhance gut health by fostering the gut colonization of beneficial bacteria and promoting the production of SCFA.
  During the pilot phase the diet is given for four weeks. Meanwhile, the intervention among pregnant mothers, the intervention is given for 20 weeks considering the nature of the availability of pregnant mothers being recruited where most of them (low risk pregnancy) were given their first clinic appointment at 16 weeks of gestational age.
  Interventions: Behavioral: Traditional Asian Diet

INTERVENTIONS:
Behavioral: Traditional Asian Diet — The personalized traditional Asian diet will be formulated based on dietary components of a typical Asian diet characterized by high intake of fruits and vegetables, whole grains, legumes, nuts, seeds, soy foods and herbs and spices; moderate intake of fish, poultry, eggs, healthy cooking oils, yogurt or functional foods and low intake of meats and sweets (Ismail et al., 2020). The diet design also considering the recommendation of personalized dietary approach by including the element of individual preferences, requirement, cultural preferences, affordability and foods availability to facilitate the adherence and response to the diet.
  Arms: Traditional Asian Diet

SUMMARY:
The research aims to elucidate a specially-designed personalized diet based on Traditional Asian Diet and its efficacy in increasing the gut colonization of Prevotella sp. and butyrate levels in pregnant mothers and the benefits in reducing infant's food allergy development.

DETAILED DESCRIPTION:
A preliminary pilot study is first will be conducted among a group of healthy volunteers. This pilot study aims to assess the feasibility of the intervention and obtain pre-eliminary data on its efficacy before proceeding to the full-scale research study. Next, in the actual trial among pregnant mothers, participants will be informed about the study and potential risk. All patients giving written informed consent will go one week screening period to assess for study eligibility prior to enrollment. At week 0, single-blind randomization (subject and health care providers except for principal investigator) will be conducted and participant will be randomized into two groups namely; the control group and the intervention group. The control group will receive standard dietary counselling on a healthy pregnancy diet. Meanwhile, the intervention group will receive dietary intervention which is tailored to the study objective to increase targeted bacteria of Prevotella sp and the short-chain fatty acids namely butyrate. The trial will be in 20 weeks duration during pregnancy and additional 12-months follow up for the delivered infants.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian and of the Malay ethnicity
* Living in Kelantan for at least 5 years
* Age 18 to 40 years
* The lower limit of ≥16th weeks and the upper limit of <20th week of gestation during enrollment to allow at least 20 weeks of dietary intervention prior to delivery. The gestational age was based on the last menstrual period (LMP) or early ultrasound examination
* Singleton pregnancy
* History of personal and family history of allergy (presence of reported or doctor-diagnosed allergic disease including asthma, eczema, food allergy, or allergy rhinitis) in participants, their partners or in their previous child or pregnancy.
* In attendance of antenatal clinic at Hospital USM or Klinik Kesihatan (Kota Bharu/Kubang Kerian/Pengkalan Chepa)
* Living area within 10 km radius of Kota Bharu, Kelantan
* Consent to participate

Exclusion Criteria:

* Significant present or having past medical history of chronic disease for example bowel, cancer disease, systemic lupus erythematosus (SLE), chronic kidney disease, heart failure, stroke, haematological malignancy, and chronic obstructive pulmonary disease.
* Significant psychiatric history including major depression and other psychotic disorders.
* Significant present or past surgical history including bowel surgeries
* Significant presence of doctor-diagnosed short intestinal bacteria overgrowth (SIBO).
* Taking any medications which may disturb the gut microbiota or intestinal function, for example, antibiotics for the past 3 months, immunosuppressive drugs, opiates, anticoagulants and etc.
* Those who plan to move out from Kelantan after delivery which may affect the follow-up.
* Those who follow a vegetarian diet will also be excluded from participating.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 92 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Maternal gut microbiome composition before and after intervention | 20 weeks
  Maternal stool samples will be collected at three pre-determined intervals (baseline (week 16), week-28 and week-36 gestation. The gut microbiota composition will be examined using the 16s rRNA sequencing. The alpha (Shannon, Simpson and Evenness Indices) and beta diversity of the gut microbiota will be compared within and between groups.
Maternal stool metabolome concentration of short chain fatty acids (SCFA) before and after intervention | 20 weeks
  Maternal stool samples will be collected at three pre-determined intervals (baseline (week 16), week-28 and week-36 gestation. The changes in stool SCFA concentration in (umol/g) will analyzed using the gas chromatography - mass spectrometry (GC-MS). The concentration (umol/g) be compared within and between groups.
Incidence of allergy development in the delivered infants and its correlation with maternal gut microbiome during pregnancy. | 12 months
  Symptoms perceived by parents/caregivers will be asked during postnatal follow-ups at day day-28, 3, 6 and 12 months of age using a validated questionnaire, the Comprehensive Early Childhood Allergy Questionnaire (CECAQ) (Minasyan A. et al.,2015). The results are then correlated with the maternal gut microbiome composition during pregnancy which was first being examined through the 16S rRNA sequencing analysis.
Incidence of allergy development in the delivered infants and its correlation with maternal stool metabolome during pregnancy. | 12 months
  Symptoms perceived by parents/caregivers will be asked during postnatal follow-ups at day day-28, 3, 6 and 12 months of age using a validated questionnaire, the Comprehensive Early Childhood Allergy Questionnaire (CECAQ) (Minasyan A. et al.,2015). The results are then correlated with the maternal gut microbiome composition during pregnancy which was first being examined through the 16S rRNA sequencing analysis.

SECONDARY OUTCOMES:
Infant's gut microbiome composition at neonatal age and its correlation with allergy development | 12 months
  Infant's stool samples collected during the neonatal age (day-0 to day-28 post delivery). The stool DNA will be extracted to examine the gut microbiome composition through 16s rRNA sequencing. The alpha (Shannon, Simpson and Evenness Indices) and beta diversity of the gut microbiota will be correlate with the incidence of allergy.
Infant's stool metabolome of the short-chain fatty acids (SCFA) concentration during neonatal age and its correlation with allergy development | 12 months
  Infant's stool samples collected during the neonatal age (day-0 to day-28 post delivery). The stool concentration of the SCFA measured in umol/g will be analyzed using the gas chromatography-mass spectrometry (GC-MS). The concentration of the SCFA (in umol/g) will be correlate with the incidence of allergy.
Infant's immune functions and allergy development | 12 months
  Infant's immune function (measured by concentration of interleukin-10/IL-10, and transforming growth factor-beta/TGF-B). The plasma will be assayed IL-10 and transforming growth factor beta (TGF-β) using the ELISA kits following the manufacturer and the concentration measured in ng/mL. The concentrations IL-10 and TGF-Beta (ng/mL) will be further examined its correlation with allergy development in infants.
Infant's gut barrier and allergy development | 12 months
  Infant's gut barrier will be measured through the serum FABP2, a marker of intestinal integrity (Vreugdenhil et al., 2011). The plasma will be assayed using the Human FABP2 ELISA kit following manufacturer instructions. The concentration of the FABP2 measured in ng/mL will be further examined its correlation with allergy development in infants.

OTHER OUTCOMES:
The changes on gut microbiome composition in healthy volunteers before and after 4 weeks dietary intervention. | 4 weeks
  Stool samples will be collected at three pre-determined intervals (baseline, week-2 and week-4) during study period. The gut microbiota composition will be examined using the 16s rRNA sequencing. The alpha (Shannon, Simpson and Evenness Indices) and beta diversity of the gut microbiota will be compared within and between groups.
The changes on stool metabolome of shiort chain fatty cids (SCFA) composition in healthy volunteers before and after 4 weeks dietary intervention. | 4 weeks
  Stool samples will be collected at three pre-determined intervals (baseline, week-2 and week-4) during study period. The stool SCFA concentration in (umol/g) will analyzed using the gas chromatography - mass spectrometry (GC-MS). The changes in SCFA concentration (umol/g) be compared within and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: NUR-FAZIMAH SAHRAN, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Derived] Sahran NF, Chong CW, Ismail IH, Taib F, Hoo PS, Palanisamy UD, Sundralingam U, Teh CSJ, Kong ZX, Ayub Q, Yoke Ling F, Hazlan SNH, Azlan M, Abdul Razak S, Tengku Din TADA, Abdullah N, Tagiling N, Tee V, Ehab Ayad M, Zheng FM, El-Omar E, Lee YY. Effects of Traditional Asian Diet on dietary fibre requirement, gut microbiome composition, and faecal and urine metabolomes in healthy Asian women: a pilot study. Benef Microbes. 2025 Apr 22:1-14. doi: 10.1163/18762891-bja00074. Online ahead of print. PMID 40312033